CLINICAL TRIAL: NCT03307109
Title: Quality of Life in Patients Having a Prosthetic Joint Infection
Acronym: QuaVIPA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0419
Record Dates: First submitted 2017-10-04; First posted 2017-10-11 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Quality of Life; Prosthetic Joint Infection
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having prosthetic joint infection: The primary aim is to measure the evolution of quality of life in patients having prosthetic joint infection during their medical care and possibly psychologic assistance in the Infectious and Tropical Diseases Department of Croix-Rousse Hospital.
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — Patients will complete two EQ-5D-5L and EQ-5D-3L quality of life questionnaires and will complete an analog visual scale during each of their follow-up visits to the Infectious and Tropical Diseases Department of Croix-Rousse hospital. No visits will be added to complete the questionnaires.

SUMMARY:
Bone and joint infections (BJI) are rare serious pathology which can lead to a very heavy handicap and sometimes to the life threatening. These are devastating diseases whose diagnosis is difficult. They are known to be associated with high mortality rates (5%) and significant morbidities responsible for functional sequelae (40% of patients) with an individual cost (prolonged hospitalization, altered quality of life) and societal (work stoppage, partial or total disability, temporary or permanent) extremely high.

These bone and joint infections have a significant impact on the quality of life of those affected who, in addition to their infection, are reduced in their autonomy and often need to be taken care of outside their home, sometimes away from home.

To the knowledge of investigators, there are few studies on the measurement of quality of life in patients with osteoarticular infection.

The aim of this study is to implement the EQ-5D-3L validated quality of life questionnaire and the EVA scale (created by EuroQol Group) for each patient with a prosthetic joint infection (IPA) on prosthesis during their medical care in the department of Infectious and Tropical Diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient having prosthetic joint infection
* Patient who did not object to participate in the study
* Patients over 18 years of age

Exclusion Criteria:

* Patient with additional psychological or psychiatric support outside the service.
* Patient benefiting from a system of legal protection (safeguard of justice, guardianship, curatorship)
* Patient participating in another study on measuring quality of life
* Patients with cognitive impairment to understand the questionnaire
* Impossibility of giving the patient informed information
* Patients with no infection diseases follow up at the CROIX ROUSSE hospital
* Patients with amputation as initial surgery for infection management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having an prosthetic joint infection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Questionnaire EQ-5D-3L | 12 to 24 months
  EQ5D is one of the most widely used health states descriptive system and has a valuation in France.
  EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 3 problem levels corresponding to patient response choices.
  A quality of life score is obtained according to the answers to the questionnaires.
Analog Visual Scale | 12 to 24 months
  Use of a Analog Visual Scale to measure the quality of life

SECONDARY OUTCOMES:
Questionnaire EQ-5D-5L | 12 to 24 months
  In the EQ-5D-5L the 5 dimensions are described by 5 problem levels corresponding to patient response choices.
  A quality of life score is obtained according to the answers to the questionnaires. In France, only the EQ-5D-3L has been validated, not yet the EQ-5D-5L which has only been translated.
  In this study investigators want compare the score obtained to the questionnaires EQ5D-5L and EQ-5D-3L to determine if EQ-5D-5L is more adapted to patients having prosthetic joint infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de reference des infections ostéo-articulaires de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No